CLINICAL TRIAL: NCT00882830
Title: Electrical Muscle Stimulation (EMS), a Preventive and Therapeutic Tool for Critical Illness Polyneuromyopathy (CIPNM)- A Randomized Controlled Parallel Intervention Trial.
Brief Title: Electrical Muscle Stimulation (EMS), a Preventive and Therapeutic Tool for Critical Illness Polyneuromyopathy (CIPNM)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Serafim Nanas, MD, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SNCT050253
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Critical Illness Polyneuromyopathy (CIPNM); ICU Acquired Weakness (ICUAW)
Keywords: ICU; myopathy; neuropathy; EMS; critical illness polyneuromyopathy; NIRS; muscle biopsy; microdialysis; CIPNM
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMS group (Experimental)
  Interventions: Procedure: EMS
- control group (No Intervention)

INTERVENTIONS:
Procedure: EMS — EMS sessions on both lower extremities (quadriceps and peroneus longus) simultaneously.
  Other Names: Electrical muscle stimulation
  Arms: EMS group

SUMMARY:
The purpose of this study is to investigate the role of EMS as a preventive and therapeutic tool of CIPNM. The investigators hypothesized that EMS will prevent the development of CIPNM or have a beneficial role as a therapeutic means in case of CIPNM appearance.

DETAILED DESCRIPTION:
CIPNM is one of the most frequent clinical problems encountered in a general ICU. Inflicted patients are characterized by generalized muscle weakness, areflexia, delayed weaning from mechanical ventilation and subsequent increased duration of ICU stay. So far, no therapeutic or preventive tool has been proposed for CIPNM.

Electrical muscle stimulation (EMS) has been proposed as an alternative exercise modality in patients with severe chronic obstructive pulmonary disease and chronic heart failure, who cannot perform active exercise. The role of EMS in ICU patients has not been evaluated so far.

We designed a randomized intervention study to assess the efficacy of EMS, as a preventive or therapeutic tool in CIPNM. The study consists of two cohorts. In the preventive cohort, patients with Apache II admission score ≥ 13, after stratified (age, gender) randomization, are assigned on the second day after admission to the EMS group or to the control group. In the observation cohort, patients with Apache II < 13 are followed clinically until interruption of sedation. Patients who regain consciousness and are cooperative are assessed clinically for CIPNM. If they are diagnosed with CIPNM, they undergo stratified randomization (age, gender, diabetes mellitus, malignancy) to EMS group or to the control group. EMS will be applied to both lower extremities of the EMS-group simultaneously (quadriceps femoris muscle and peroneus longus) on a daily basis. EMS sessions will continue until patient discharge or death. EMS sessions are supplementary to standard physiotherapy practice applied to all ICU patients.

Primary end point is the diagnosis of CIPNM. Secondary end points are 1) the duration of weaning from the ventilator, 2) time to ICU discharge, 3) muscle mass preservation, 4) muscle strength, 5) muscle properties and structure. The primary and secondary endpoints will be assessed as follows: medical research scale (MRC) for clinical evaluation of muscle strength, handgrip dynamometry, muscle mass evaluation with ultra-sonography, muscle biopsies, maximal inspiratory pressure, tissue oxygen saturation assessed with near infrared spectroscopy (NIRS), muscle microdialysis, electromyography (EMG).

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted in ICU of Evaggelismos Hospital

Exclusion Criteria:

* age < 18 years
* pregnancy
* pre-existing neuromuscular disease (e.g. Gravis)
* connective tissue disease
* fractures or skin lesions that do not allow the implementation of EMS
* BMI > 35 kg/m2
* brain death
* terminal disease
* length of stay < 48 hours
* presence of pacemaker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of CIPNM | June 2009

SECONDARY OUTCOMES:
Duration of weaning, time to ICU discharge, muscle mass preservation, muscle strength, muscle properties and structure. | June 2011

CONTACTS AND LOCATIONS:
Overall Officials: Serafim Nanas, MD, Principal Investigator — University of Athens
Locations (1):
- First Critical Care Unit, Evaggelismos Hospital, School of Medicine, University of Athens, Athens, Greece

REFERENCES:
- [Result] Routsi C, Gerovasili V, Vasileiadis I, Karatzanos E, Pitsolis T, Tripodaki E, Markaki V, Zervakis D, Nanas S. Electrical muscle stimulation prevents critical illness polyneuromyopathy: a randomized parallel intervention trial. Crit Care. 2010;14(2):R74. doi: 10.1186/cc8987. Epub 2010 Apr 28. PMID 20426834
- [Result] Karatzanos E, Gerovasili V, Zervakis D, Tripodaki ES, Apostolou K, Vasileiadis I, Papadopoulos E, Mitsiou G, Tsimpouki D, Routsi C, Nanas S. Electrical muscle stimulation: an effective form of exercise and early mobilization to preserve muscle strength in critically ill patients. Crit Care Res Pract. 2012;2012:432752. doi: 10.1155/2012/432752. Epub 2012 Apr 1. PMID 22545212
- [Result] Gerovasili V, Stefanidis K, Vitzilaios K, Karatzanos E, Politis P, Koroneos A, Chatzimichail A, Routsi C, Roussos C, Nanas S. Electrical muscle stimulation preserves the muscle mass of critically ill patients: a randomized study. Crit Care. 2009;13(5):R161. doi: 10.1186/cc8123. Epub 2009 Oct 8. PMID 19814793
- [Result] Gerovasili V, Tripodaki E, Karatzanos E, Pitsolis T, Markaki V, Zervakis D, Routsi C, Roussos C, Nanas S. Short-term systemic effect of electrical muscle stimulation in critically ill patients. Chest. 2009 Nov;136(5):1249-1256. doi: 10.1378/chest.08-2888. Epub 2009 Aug 26. PMID 19710290
- [Result] Tzanis G, Vasileiadis I, Zervakis D, Karatzanos E, Dimopoulos S, Pitsolis T, Tripodaki E, Gerovasili V, Routsi C, Nanas S. Maximum inspiratory pressure, a surrogate parameter for the assessment of ICU-acquired weakness. BMC Anesthesiol. 2011 Jun 26;11:14. doi: 10.1186/1471-2253-11-14. PMID 21703029